CLINICAL TRIAL: NCT06707168
Title: ACCURACY of DIGITAL INTRAOCULAR PRESSURE MEASUREMENT AT the END of PARS PLANA VITRECTOMY SURGERY
Brief Title: INTRAOCULAR PRESSURE MEASUREMENT AT the END of PARS PLANA VITRECTOMY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Eng, Chief of Ophthalmology, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6310
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pars Plana Vitrectomy
Keywords: intraocular pressure; pars plana vitrectomy
MeSH Terms: interventions — Digital Rectal Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgeon #1 (Other): One by digital palpation over the limbal area; and the other using a short wooden cotton-tipped applicator (CTA) over the limbal area.
  Interventions: Diagnostic Test: Digital palpation; Diagnostic Test: Cotton-tipped applicator (CTA)
- Surgeon #2 (Other): One by digital palpation over the limbal area; and the other using a short wooden cotton-tipped applicator (CTA) over the limbal area.
  Interventions: Diagnostic Test: Digital palpation; Diagnostic Test: Cotton-tipped applicator (CTA)

INTERVENTIONS:
Diagnostic Test: Digital palpation — Digital palpation for IOP measurement
Diagnostic Test: Cotton-tipped applicator (CTA) — Cotton-tipped applicator (CTA) for IOP measurement

SUMMARY:
Intraocular pressure is measured regularly at any and all visits with your eye doctor or optometrist.

The purpose of this study is to compare measurements of eye pressure at the end of the surgery, comparing the ability of a gloved finger or sterile cotton-tipped applicator ("Q-tip") to accurately measure intraocular pressure against a standardized instrument designed for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing Pars Plana Vitrectomy between June 25, 2024 - and December 30, 2024, will be included.
2. Patients aged 18 years or older
3. Patients able to give informed consent

Exclusion Criteria:

1. Patients with complicated Pars Plana Vitrectomy (choroidal hemorrhage, retrobulbar hemorrhage)
2. Patients with irregular cornea surface will be excluded (keratoconus, band keratopathy, corneal edema, corneal transplant, cornea scarring)
3. Patients undergoing combined scleral buckling at time of surgery
4. Patients with previous glaucoma filtration surgery (ie. trabeculectomy or tube shunt surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure measurement | From enrolment to end of treatment at 8 weeks
  Intraocular pressure accuracy between surgeons' estimate and tonometer IOP measurement.

SECONDARY OUTCOMES:
Intraocular pressure measuring agreement | From enrolment to end of treatment at 8 weeks
  1. Intraocular pressure surgeon measuring agreement with digital palpation.
  2. Intraocular pressure surgeon measuring agreement with short wooden stick cotton swab.

IPD SHARING:
Plan to Share IPD: No
No identifying information will be shared

REFERENCES:
- [Background] Acar N, Kapran Z, Unver YB, Altan T, Ozdogan S. Early postoperative hypotony after 25-gauge sutureless vitrectomy with straight incisions. Retina. 2008 Apr;28(4):545-52. doi: 10.1097/IAE.0b013e318162b008. PMID 18398355
- [Background] Wilde C, Bhardwaj P, King A, Kumudhan D, Foss A, Orr G, Zaman A. First postoperative day review in eyes undergoing pars plana vitrectomy, encirclement and endotamponade to check intraocular pressure: Is it necessary? Int Ophthalmol. 2020 Oct;40(10):2577-2583. doi: 10.1007/s10792-020-01438-w. Epub 2020 Jun 1. PMID 32488595
- [Background] Alexander P, Michaels L, Newsom R. Is day-1 postoperative review necessary after pars plana vitrectomy? Eye (Lond). 2015 Nov;29(11):1489-94. doi: 10.1038/eye.2015.134. Epub 2015 Aug 28. PMID 26315702